CLINICAL TRIAL: NCT00145262
Title: Therapeutic Angiogenesis Using Cell Transplantation (TACT) Study at Nagoya
Brief Title: TACT-NAGOYA: Therapeutic Angiogenesis Using Cell Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Other Study IDs: 66
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-12-30 (Estimated); Status verified 2003-08

CONDITIONS: Buerger Disease; Arteriosclerosis Obliterans
Keywords: critical limb ischemia; bone marrow mononuclear cells; angiogenesis; vasculogenesis; Arteriosclerosis Obliterans (ASO); Ischemic ulcers
MeSH Terms: conditions — Thromboangiitis Obliterans; Arteriosclerosis Obliterans; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Autologous Bone Marrow Mononuclear Cell Implantation

SUMMARY:
Clinical studies have established that implantation of bone marrow mononuclear cells (BM-MNCs) or peripheral blood mononuclear cells (PB-MNCs) into ischaemic limbs increases collateral vessel formation. We, the investigators at Nagoya University, further investigated the efficacy and safety of autologous implantation of BM-MNCs or PB-MNCs in patients with severe ischaemic limbs who have no other alternative therapeutic options. We also examined a potential limiting factor which reduced the efficacy of therapeutic angiogenesis using cell transplantation (TACT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have chronic limb ischemia, including rest pain, non-healing ischemic ulcers, or both, and who are not candidates for nonsurgical or surgical revascularisation.

Exclusion Criteria:

* Poorly controlled diabetes mellitus (hemoglobin A1c [HbA1c] > 6.5% and proliferative retinopathy)
* Evidence of malignant disorder during the past 5 years
* Subjects who cannot survive more than 1 year with other complications
* Malignant rheumatic arthritis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Toyoaki Murohara, MD, PhD, Principal Investigator — Department of Cardiology, Nagoya University Graduate School of Medicine
Locations (1):
- Department of Cardiology, Nagoya University Graduate School of Medicine, Nagoya, Japan

REFERENCES:
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Derived] Kajiguchi M, Kondo T, Izawa H, Kobayashi M, Yamamoto K, Shintani S, Numaguchi Y, Naoe T, Takamatsu J, Komori K, Murohara T. Safety and efficacy of autologous progenitor cell transplantation for therapeutic angiogenesis in patients with critical limb ischemia. Circ J. 2007 Feb;71(2):196-201. doi: 10.1253/circj.71.196. PMID 17251666